CLINICAL TRIAL: NCT05455528
Title: Preoperative Renal Insufficiency Predicts Postoperative Adverse Outcomes: A Matched Cohort Study Using the NSQIP Database
Brief Title: Preoperative Renal Insufficiency Predicts Postoperative Adverse Outcomes
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chao-Shun Lin, principal investigator, Taipei Medical University Hospital
Other Study IDs: 202206019
Record Dates: First submitted 2022-07-03; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Renal Insufficiency; Morality
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- renal insufficiency group: 1. Surgical population currently on dialysis
  2. Surgical population with estimated GFR < 60 ml/min per 1.73 square meter within 90days before the index surgery. The estimated GFR
  Interventions: Diagnostic Test: estimated GFR calculation
- Non-renal insufficiency group: Defined as the study subjects with eGFR > 90 60 ml/min per 1.73 square meter within 90 days before the index surgery
  Interventions: Diagnostic Test: estimated GFR calculation

INTERVENTIONS:
Diagnostic Test: estimated GFR calculation — The estimated GFR is computed with Modification of Diet in Renal Disease (MDRD) formula

SUMMARY:
The main purpose of this study is to evaluate the risk of postoperative mortality and complications in surgical populations with preoperative renal insufficiency.

DETAILED DESCRIPTION:
This retrospective cohort study use the National Surgical Quality Improvement Program (NSQIP) database to evaluate the risk of postoperative morbidity and mortality in the surgical population. Patients with estimated. glomerular filtration rate(GFR) < 60 ml/min per 1.73 square meter are defined as the renal insufficiency group. Patients with estimated GFR > 90 ml/min per 1.73 square meter are defined as patients without renal insufficiency. Propensity score-matching methods and multivariate logistic regression are used to calculate the risk of postoperative morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with estimated GFR < 60 ml/min per 1.73 square meter or currently on dialysis are included in renal insufficiency group.
* Patients with estimated GFR > 90 ml/min per 1.73 square meter are included in non-renal insufficiency group

Exclusion Criteria:

* Patients population with estimated GFR between 60-90 is not included in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study analyze surgical patient data from the American College of SurgeonsNational Surgical Quality Improvement Program (ACS-NSQIP) that was acquired between 2013 and 2018.
Sampling Method: Non-Probability Sample
Enrollment: 2421286 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Risk of postoperative mortality | 30 days after surgery date
  Calculate risk of postoperative 30-day in-hospital mortality between groups

SECONDARY OUTCOMES:
Risk of postoperative morbidities | 30 days after surgery date
  Postoperative events, including pneumonia, septic shock, stroke, deep vein thrombosis/thrombophlebitis, myocardial infarction and postoperative bleeding are included

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Shun Lin, MD, PhD, Study Chair — Department of Anesthesiology, Taipei Medical University Hospital, 252 Wuxing St., Taipei 110 Taiwan
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan ( R.o.c.), Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liao YC, Chang CC, Chen CY, Liu CC, Liao CC, Shih YV, Lin CS. Preoperative renal insufficiency predicts postoperative adverse outcomes in a mixed surgical population: a retrospective matched cohort study using the NSQIP database. Int J Surg. 2023 Apr 1;109(4):752-759. doi: 10.1097/JS9.0000000000000278. PMID 36974714